CLINICAL TRIAL: NCT02719015
Title: Phase I/II Dose Escalation and Cohort Expansion of Safety and Tolerability Study of Intratumoral rAd.CD40L (ISF35) in Combination of Systemic Pembrolizumab in Patients With Refractory Metastatic Melanoma
Brief Title: Dose Escalation and Cohort Expansion of Safety and Tolerability Study of Intratumoral rAd.CD40L (ISF35) in Combination of Systemic Pembrolizumab in Patients With Refractory Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No IND Serial #
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Memgen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0199
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Melanoma
Keywords: Melanoma; Refractory Metastatic Melanoma; rAd.CD40L; ISF35; Intratumoral; IT; Pembrolizumab; Keytruda; MK-3475; SCH-900475; MM
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rAd.CD40L + Pembrolizumab (Experimental): The dose escalation phase will include rAd.CD40L dose escalation and increase in the number of injected sites/lesions. Once patients tolerate dose level 1 (1 injection site and 1x1011vp-MTD) in Dose Escalation cohort, Expansion cohort will open with same maximum number of injection sites at maximum tolerated dose from Dose Escalation cohort.
  All participants receive same dosage of Pembrolizumab in both phases.
  Interventions: Drug: rAd.CD40L; Drug: Pembrolizumab

INTERVENTIONS:
Drug: rAd.CD40L — Dose Escalation Phase Starting Dose: 5x10^10 vp per tumor as an injection directly into 1-3 tumors every 3 weeks. Same tumors injected for each of the 4 injections at week 0, 3, 6 and 9. If the dose well tolerated, the rAd.CD40L escalated to 1x10^11 vp. Subsequently enrolled patients injected at the same dose of 1x10^11 vp. Number of injected sites/tumors increased to two sites/lesions if patients have >/=2 injectable lesions, at the same injection dose of 1x10^10 up to three separate sites/lesions if patients have > 3 injectable lesions.
  Dose Expansion Phase Starting Dose: MTD from Dose Escalation Phase.
  Other Names: ISF35
Drug: Pembrolizumab — Dose Escalation and Expansion Phases: 2 mg/kg by vein every 3 weeks.
  Other Names: Keytruda; MK-3475; SCH-900475

SUMMARY:
The goal of this clinical research study is to find the highest tolerated dose of rAd.CD40L (also called ISF35) when given with pembrolizumab to patients with melanoma. Researchers also want to learn if the highest tolerated dose of ISF35 and pembrolizumab can help to control the disease.

The safety of this drug combination will be also be studied.

DETAILED DESCRIPTION:
Study Groups:

If participant is found to be eligible to take part in this study, they will be assigned to 1 of 2 dose levels of ISF35 based on when they join this study. Up to 6 participants will be enrolled in the first group and up to 24 participants will be enrolled in the second group. The first group of participants will receive the lowest dose level. If no intolerable side effects are seen, all other participants enrolled in the study will receive the highest dose. If participant is assigned to the first group, they will not be able to move up to the second group.

All participants will also receive the same dose of pembrolizumab.

Study Drug Administration:

Participants will receive ISF35 as an injection directly into 1-3 tumors every 3 weeks. The injections will be done in the clinic or at the interventional radiology suite. The study staff may use image guidance such as ultrasound, CT, and/or MRI to help inject the drug into the tumor.

Participants will also receive pembrolizumab by vein over about 30 minutes every 3 weeks.

Study Visits:

At Week 0 (the first week participants receive treatment):

* Participant will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and to check participant's immune system.
* Participant will have a tumor biopsy to check how the disease is responding to the study drug. To collect a biopsy, the area of skin is numbed with anesthetic and a small cut is made to remove all or part of the affected tissue. This biopsy will be performed within 24 hours of the first dose.
* The tumors will be photographed and measured. For the photographs, participant's private areas will be covered (as much as possible), and a picture of their face will not be taken unless there are tumors on their face.

At Weeks 1 and 2:

* Participant will have a physical exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.

At Weeks 3, 6, and 9 (± 3 days):

* Participant will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and to check participant's immune system.
* During Week 6 only, participant will have a biopsy of 1 of the tumors that has been injected with the study drug and 1 of the tumors that they did not have an injection in to learn if the tumors have responded to the study drug. Researchers also want to learn if participant has any genetic mutations (changes) that may change how they respond to the study drug. The tumors will also be photographed and measured.

Length of Study:

Participant may receive the study drugs for up to 9 weeks. Participant will be taken off study if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation on the study will be over after about 2 years of follow-up visits.

End-of-Study Visit:

About 3 weeks after participant's last dose of study drug (Week 12) or as soon as they stop taking the study drug (if they stop taking the study drug before Week 9):

* Participant will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests, to check participant's immune system, and to learn if the study drug has had any effect on the disease.
* Participant will have an MRI, CT, or positron emission computed tomography (PET)/CT scan and the tumors will be photographed and measured.

Follow-Up

Within 2 weeks after participant's last dose of study drugs and then every 8-12 weeks after that for up to 2 years:

* Participant will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests, to check participant's immune system, and to learn if the study drug has had any effect on the disease.
* Participant will have MRI, CT, and/or PET/CT scans to check the status of the disease. The tumors will also be measured and photographed. Participant's doctor will decide what type of scans they will have.
* At participant's first follow-up visit after they stop taking the study drug, they will have a tumor biopsy to check the status of the disease.

If participant chooses to receive care at another hospital, the study staff will call them every 3 months for up to 2 years after their last dose of study drugs to learn how they are doing. The calls should last about 5 minutes.

This is an investigational study. ISF35 is not FDA approved or commercially available. It is currently being used for research purposes. Pembrolizumab is FDA approved and commercially available for the treatment of melanoma and non-small cell lung cancer (NSCLC). The study doctor can explain how the study drugs are designed to work.

Up to 36 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Dose escalation: Patients with metastatic melanoma with measurable, stage III (in transit lesions) or stage IVA, IVB or IVC disease (at least 2 measurable lesions/tumors. Patients will be required to have one more lesion present than the number the current dose level requires since one lesion will be left untreated.
2. Expansion cohorts: Patients with metastatic melanoma with measurable, stage III (in transit lesions) or stage IVA, IVB or IVC disease at least two measurable lesions/tumors
3. Patients who have tested positive for a BRAF mutation may have received prior BRAF inhibitor therapy as a prior line of systemic therapy. Patients may have received up to 2 prior lines of therapy with a checkpoint inhibitor (CPI), which may have included pembrolizumab, nivolumab, or ipilimumab. These agents may have been administered as single-agent treatment, in combination with each other, or in combination with other agents. Patients who have received prior treatment with ipilimumab must have relapsed after achieving a response to prior ipilimumab treatment. This response may have been achieved with ipilimumab administered as single-agent therapy or in combination with another treatment. Patients who have received prior treatment with pembrolizumab or nivolumab must have progression of disease after at least 4 doses of either drug alone or in combination with other agents.
4. Age >/= 18 years
5. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 - 1 within 30 days of signing informed consent.
6. Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
7. Platelet count greater than or equal to 100,000/mm3
8. white blood cell count (WBC) >/=3000/mm3
9. Serum ALT and AST <3 the upper limit of normal (ULN); <5 ULN if there is liver involvement secondary to the tumor
10. Serum creatinine </= 2.0 mg/dl
11. Seronegative for HIV antibody
12. Patients with a negative pregnancy test (urine or serum) must be documented within 14 days of screening for women of childbearing potential (WOCBP). A WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e. who has not had menses at any time in the preceding 12 consecutive months).
13. Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), the patient agrees to continue to use a barrier method of contraception throughout the study such as: condom, diaphragm, hormonal, intrauterine device (IUD), or sponge plus spermicide. Abstinence is an acceptable form of birth control.

Exclusion Criteria:

1. Patients who have previously received anti cluster of designation antigen 40 (CD40) (Agonistic) therapy prior Adjuvant Interferon (IFN-α), is allowed if last dose was received at least 6 months from enrolling to protocol.
2. Active autoimmune disease requiring disease modifying therapy.
3. Concurrent systemic steroid therapy higher than physiologic dose (>7.5 mg/Day of prednisone).
4. Any form of active primary or secondary immunodeficiency.
5. Prior malignancy except the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, thyroid cancer (except anaplastic) or any cancer from which the patient has been disease-free for 2 years.
6. Subjects who have received prior oncolytic therapy or prior therapy with and TLR agonist including topical agents. Subjects that have received experimental vaccines or other immune therapies should be discussed with the medical monitor or the Principal Investigator (PI) to confirm eligibility.
7. Active systemic infections requiring intravenous antibiotics.
8. Prior systemic therapy, radiation therapy, or surgery within 28 days of starting study treatment. Palliative radiotherapy to a limited field or palliative cryoablation is allowed after consultation with the principle Investigator, at any time during the study participation including screening.
9. Patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Intratumoral rAd.CD40L | 3 weeks
  MTD defined as the dose with the smallest absolute difference between the estimate of pi and the true pT for which Prob (pi > pT | data) is less than 5%.
Overall Response Rate (ORR) of Intratumoral rAd.CD40L | 12 weeks
  Tumor response to therapy assessed using immune-related response criteria (irRC), which is a modified version of the World Health Organization (WHO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Diab, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org